CLINICAL TRIAL: NCT03789422
Title: Efficacy and Safety of Levocetirizine Alone or in Combination With Tranexamic Acid in the Treatment of Spontaneous Chronic Urticaria. Multicentric Controlled Randomized Study in Cross-over, Double-blind
Brief Title: Tranexamic Acid and Spontaneous Chronic Urticaria
Acronym: TACUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TACUS- 38RC18.103
Record Dates: First submitted 2018-10-17; First posted 2018-12-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Multicentric controlled randomized crossover study, double-blind
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Association drugs (Active Comparator): levocetirizine 10mg/day + tranexamic acid (AT) 2g/day for a month
  Interventions: Drug: association of levocetirizine and tranexamic acid
- one drug (Active Comparator): Levocetirizine 20 mg/day for a month
  Interventions: Drug: Levocetirizine only

INTERVENTIONS:
Drug: association of levocetirizine and tranexamic acid — levocetirizine 10 mg/day + tranexamic acid 2 g/day
  Arms: Association drugs
Drug: Levocetirizine only — levocetirizine 20 mg/day
  Arms: one drug

SUMMARY:
Spontaneous chronic urticaria (UCS) is a disease that affects 1% of the general population with a potentially severe impact on quality of life. Most patients respond favorably to long-term antihistamine treatment, but sometimes it is necessary to give a high dose (4 times the formal dose, Berlin consensus 2016). These high doses are often accompanied by side effects requiring cessation of treatment. The therapeutic alternative is then omalizumab, an expensive biotherapy. UCS is secondary to non-specific mast cell activation. It has been shown to be associated with activation of fibrinolysis that correlates with the severity of symptoms. Patients with UCS resistant to levocetirizine were shown to have higher D-dimer levels than patients who responded to antihistamines. Tranexamic acid is a molecule with antifibrinolytic propertiesSeveral cases of severe chronic urticaria responding favorably to treatment with tranexamic acid have been reported. In our department, Investigators also noticed the improvement of some of their patients on tranexamic acid. The combination of these two treatments appears to be synergistic: action on histamine receptors and control of fibrinolysis.

The investigators propose to evaluate the association of tranexamic acid and levocetirizine for the treatment of chronic spontaneous urticaria.

DETAILED DESCRIPTION:
Multicentric controlled randomized crossover study, double-blind To evaluate the efficacy and safety of levocetirizine 10mg / day + tranexamic acid (AT) 2g / day versus levocetirizine 20mg / day alone in the chronic treatment of chronic urticaria evaluated at 4 weeks.

A hierarchical analysis will be implemented in the following order:

1. Non-inferiority of the combination levocetirizine 10 mg / day + tranexamic acid (TA) 2 g / day versus levocetirizine alone 20 mg / day in terms of effectiveness
2. Superiority of the combination levocetirizine 10 mg / day + tranexamic acid (AT) 2 g / day versus levocetirizine alone 20 mg / day in terms of tolerance
3. Superiority of levocetirizine 10mg / day + tranexamic acid (AT) 2g / day versus levocetirizine alone 20mg / day in terms of effectiveness Each objective will be tested sequentially if and only if the previous objective is validated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous chronic urticaria, according to the criteria of the European Academy of Allergology and Clinical Immunology (EAACI) in agreement with the European Dermatology Forum (EDF), and the World Allergy Organization (WAO), corresponding to an association of the following symptoms : urticarial eruptions and / or recurrent angioedema for at least 6 weeks

Exclusion Criteria:

* Urticaria associated with a specific systemic disease including cutaneous and systemic mastocytosis, urticarial vasculitis, autoinflammatory diseases associated with cryopyrin
* Bradykinin angioedema and isolated angioedema whose origin is not clearly attributable to spontaneous chronic urticaria.
* Presence of a contraindication to tranexamic acid and to levocetirizine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evolution of the Urticaria Activity Score 7 (UAS7) | 28 days
  Evolution of the UAS7 score between the beginning (J0) and the end (J28) of the treatment period. To calculate the score, the patient rates the number of papules and itching intensity from 0 to 3 daily for 7 days. 0 corresponds to no papules and no itching, 3 corresponds to more than 50 papules per 24h and intense itching that can cause daily life. This makes a score of 0 to 6 per day accumulated over 7 days, ranging from 0 to 42.
Tolerance of the association tranexamic acid and levocetirizine | 28 days
  Number of adverse events

SECONDARY OUTCOMES:
To demonstrate the non-inferiority of levocetirizine 10mg / day + tranexamic acid (AT) 2g / day versus levocetirizine alone 20mg / day in terms of efficacy on the Angioedema Activity Score (AAS) | 28 days
  Evolution of the AAS score between the beginning (J0) and the end (J28) of the end of treatment. The AAS score is a The AAS consists of 5 questions as well as an opening question. A score between 0 and 3 is assigned to every answer field. The question scores are summed up to an AAS day sum score, 7 AAS day sum scores to an AAS week sum score (AAS7). Accordingly, the minimum and maximum possible AAS scores are 0-15 (AAS day sum score), 0-105 (AAS7).
Clinical characteristics of responders | 28 days
  Identify the clinical characteristics of responders to the combination rather than antihistamines alone.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence BOUILLET, PhD, Principal Investigator — Internal Medicine - University Hospital Grenoble-Alpes
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France